CLINICAL TRIAL: NCT07113314
Title: Phase II Study for Prophylaxis of Febrile Neutropenia by Supplementation With Lactoferrin in Oncohematologic Children Undergoing High-intensity Chemotherapy Treatment
Brief Title: Prophylaxis of Febrile Neutropenia With Lactoferrin in Oncohematologic Children Undergoing Induction Chemotherapy
Acronym: Lactoferrin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Marco Zecca, Principal Investigator, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Lactoferrin 3527/2016
Record Dates: First submitted 2025-07-14; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Febrile Neutropenia (FN); Sepsis; Chemotherapy Treatment
Keywords: chemotherapy treatment; Sepsis; Febbrile neutropenia
MeSH Terms: conditions — Febrile Neutropenia; Sepsis

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled study
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lactoferrin (Experimental): Patients in the prophylaxis group will receive, in addition to standard treatment, a orodispersible formulation of bovine lactoferrin or bLF (Mosiac®) at the standard dose of 200 mg/day, in single administration, from the start of chemotherapy treatment and for the duration of the risk period.
  Interventions: Dietary Supplement: Lactoferrin Bovine
- Placebo (Placebo Comparator): Patients in the control group will receive only the standard treatment provided by their clinical center with placebo added from the start of chemo/radiotherapy treatment and throughout the duration of the risk period.
  Interventions: Dietary Supplement: Lactoferrin Bovine

INTERVENTIONS:
Dietary Supplement: Lactoferrin Bovine — In addition to standard treatment, a gold-soluble formulation of bovine lactoferrin or bLF (Mosiac®) at the standard dose of 200 mg/day, in single administration, from the start of chemo/radiotherapy treatment and throughout the risk period.

SUMMARY:
Test, in a randomized phase II trial, the safety and efficacy of lactoferrin prophylaxis in preventing the occurrence of febrile neutropenia and sepsis, with particular regard to forms due to multidrug-resistant Gram-negative bacteria.

ELIGIBILITY:
Inclusion Criteria:

Patients with severe neutropenia lasting >7 days:

* non-High Risk Acute Lymphoblastic Leukemia ( ALL) under induction treatment
* Acute Myeloid Leukemia (AML) (first two cycles of treatment)
* B cell - non Hodgkin Lymphoma (NHL) Ability to take oral lactoferrin therapy and perform the diagnostic tests established by the protocol

Exclusion Criteria:

* Previous chemotherapy treatments
* Past history of colonization/infection by multidrug-resistant pathogens
* Inability to take LF by mouth
* Refusal to participate in the study

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 160 (Actual)
Dates: Start 2016-10-06 (Actual); Primary Completion 2018-03-03 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Primary Outcome | From treatment up to 90 days
  Presence or absence of febrile neutropenia or sepsis

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo Pavia, Pavia, Italy, Italy